CLINICAL TRIAL: NCT03091127
Title: Real-world Use of Carfilzomib Among Multiple Myeloma Patients in Europe Who Have Received at Least One Prior Therapy.
Brief Title: Real-world Use of Carfilzomib Among Multiple Myeloma Patients in Europe
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20150262
Record Dates: First submitted 2017-01-30; First posted 2017-03-27 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the recent addition of carfilzomib as a treatment option for multiple myeloma, no data is available yet on how the drug is being used outside of the clinical trial setting.

This study will therefore provide essential data to demonstrate the real world utilization of carfilzomib in routine clinical practice, including dosage, administration schedule, regimen, duration of treatment and reason for discontinuation in Europe.

DETAILED DESCRIPTION:
With the recent addition of carfilzomib as a treatment option for multiple myeloma, no data is available yet on how the drug is being used outside of the clinical trial setting.

The Primary Objective is to describe carfilzomib utilisation in routine clinical practice, including dosage, administration schedule, regimen, duration of treatment and reason for discontinuation.

* Secondary Objectives:
* Describe the population treated with carfilzomib in terms of demographics, multiple myeloma (MM) disease characteristics, treatment history, and comorbidities.
* Describe the safety profile of carfilzomib in routine clinical practice.
* Describe response to treatment as assessed by the physician and recorded in the medical file.
* Describe healthcare resource utilisation of subjects treated with carfilzomib, in terms of unplanned hospitalisations.
* Describe the reasons for choosing carfilzomib as the MM treatment of choice.
* Describe specific concomitant therapy (bisphosphonates, thromboprophylaxis, antihypertensive treatment, anti-infective treatment) and whether these therapies were used as prophylaxis or as treatment.
* Describe a cardiovascular assessment at carfilzomib regimen initiation and at occurrence of cardiac adverse events, where available per routine care (electrocardiogram [ECG], echocardiography, left ventricular ejection fraction).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of carfilzomib initiation
* At least one prior line of MM treatment has been received
* Carfilzomib treatment has been initiated per routine practice and is currently ongoing
* At least one administration of carfilzomib in a combination regimen (ie, not monotherapy) has been received
* Provided written informed consent prior to abstraction of any data, in countries where written informed consent is required.
* Subjects who previously completed treatment with carfilzomib in a clinical trial, a compassionate use program or through routine practice, are eligible to take part in the study.
* Subjects who receive radiotherapy concurrently with carfilzomib treatment are also eligible to take part in the study.
* Subjects who initiate carfilzomib treatment on a combination regimen, subsequently discontinue all concomitant medications but remain on carfilzomib monotherapy in later cycles, remain eligible for participation in the study.
* Subjects who are also enrolled in other observational studies in which standard of care is not altered are eligible to take part in the study,

Exclusion Criteria:

* Subjects who are enrolled in a carfilzomib clinical trial will not be eligible to additionally take part in this observational study.
* Subjects who are receiving carfilzomib treatment within a compassionate use program will not be eligible to take part in this observational study. If a subject who has enrolled into this observational study, also enrolls in a clinical trial in which MM treatment and/or disease management is protocol-specified, the subject becomes ineligible and the subject's data will be censored from the time the subject enrolled the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Myeloma
Sampling Method: Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Carfilzomib starting dose | 18 months
  Carfilzomib dose at first administration
Carfilzomib dose | 18 months
  Carfilzomib dose at subsequent administrations
Carfilzomib dose modification | 18 months
  Modification includes change in dose level, dose interruption, and dose delays
Time to carfilzomib dose modification | 18 months
  At least one carfilzomib dose modification, escalation or reduction
Reason for dose modification | 18 months
  Reason for dose modification or delay
Number of cycles started | 18 months
  Number of carfilzomib treatment cycles started throughout study period
Carfilzomib regimen | 18 months
  Treatment combination
Carfilzomib dosing frequency | 18 months
  Number of administrations per cycle
Carfilzomib dosing schedule | 18 months
  Timing of carfilzomib administration within treatment cycle
Carfilzomib duration of treatment | 18 months
  Duration of carfilzomib treatment
Starting dose of concomitant anti-myeloma agents | 18 months
  Dose of combination agents (e.g. lenalidomide or dexamethasone) at baseline
Dose modification for concomitant anti-myeloma agents | 18 months
  Modification includes change in dose level, dose interruption, and dose delays
Reason for frequency modification | 18 months
  At least 1 change in frequency of carfilzomib administration.
Reason for change in frequency of concomitant multiple myeloma therapies | 18 months
  Reason for change in frequency of administration.

SECONDARY OUTCOMES:
International Staging System (ISS) score and revised ISS stage at diagnosis and carfilzomib regimen initation | 18 months
  International Staging System (ISS) score of I, II, III, or unkown
Eastern Cooperative Oncology Group (ECOG) performance status | 18 months
  ECOG performance status category at multiple myeloma diagnosis and carfilzomib regimen initiation.
Cytogenetic risk profile at diagnosis | 18 months
  Cytogenetic risk profile at diagnosis
Presence of CRAB features (i.e. hypercalcemia, renal insufficiency, anemia and/or bone pain) | 18 months
  Presence of CRAB features at MM diagnosis
Presence of comorbidities | 18 months
  Diagnosed at any point in time before carflzomib regimen initiation
Previously received anti-myeloma treatment | 18 months
  Treatment history
Response to prior treatment | 18 months
  Response to prior treatment received before initiation of carfilzomib
Number of prior relapses | 18 months
  Type of relapse (molecular, hematologic, or symptomatic)
Adverse event | 18 months
  All grade 3 or above adverse events.
Time to adverse event | 18 months
  All grade 3 or above adverse events
Electrocardiogram (ECG) changes | 18 months
  ECG changes as recorded in tests performed per routine practice
Decrease in left ventricular ejection fraction (LVEF) | 18 months
  LVEF decrease as recorded in tests performed per routine practice
Initiation or dose increase of antihypertensive treatment | 18 months
  Initiation or dose increase of existing antihypertensive treatment
Initiation or dose increase of existing heart failure treatment | 18 months
  Initiation or dose increase of existing heart failure treatment
Response to carfilzomib treatment | 18 months
  Physician-assessed response as recorded on the medical charts
Type of relapse | 18 months
  Molecular, hematologic or symptomatic relapse
Number of unplanned hospitalisations | 18 months
  Initiation or dose increase of existing heart failure treatment
Concomitant therapy not part of the carfilzomib regimen | 18 months
  Concomitant therapy not part of the carfilzomib regimen
Planned subsequent treatment regimen | 18 months
  Planned subsequent treatment regimen catergory
Patient age | 18 months
  Patient age
Patient sex | 18 months
  Patient sex
Patient height | 18 months
  Patient height
Patient weight | 18 months
  Patient weight
MRI (magnetic resonance imaging) performed at MM diagnosis and carfilzomib regimen initiation. | 18 months
  MRI (magnetic resonance imaging)
PET-CT (positron emission tomography-computed tomography) performed at MM diagnosis and carfilzomib regimen initiation. | 18 months
  PET-CT (positron emission tomography-computed tomography)
Measurement of Serum M component at MM diagnosis and carfilzomib regimen initiation. | 18 months
  Serum M component
Measurement of Urine M component at MM diagnosis and carfilzomib regimen initiation. | 18 months
  Urine M component
Measurement of serum albumin at MM diagnosis and carfilzomib regimen initiation. | 18 months
  Serum albumin
Measurement of serum beta-2-microglobulin at MM diagnosis and carfilzomib regimen initiation. | 18 months
  Beta-2-microglobulin
Measurement of percent of plasma cells in bone marrow at MM diagnosis and carfilzomib regimen initiation. | 18 months
  Percent of plasma cells in bone marrow
Baseline measurement of lactate dehydrogenase at MM diagnosis and carfilzomib regimen initiation. | 18 months
  Lactate dehydrogenase
ECG (electrocardiogram) | 18 months
  ECG (electrocardiogram)
Echocardiogram | 18 months
  Echocardiogram
LVEF (left ventricular ejection fraction) assessment | 18 months
  LVEF (left ventricular ejection fraction) assessment
Computed Tomography (CT) performed at MM diagnosis and carfilzomib regiment initiation. | 18 Months
  Computed tomography
Myeloma/Osteolytic lesions detected by MRI, PET-CT, and X-ray at MM diagnosis and carfilzomib regimen initiation | 18 months
  Myeloma/Osteolytic lesions detected by MRI, PET-CT, and X-ray at MM diagnosis and carfilzomib regimen initiation

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (114):
- Austria (12):
  - Krankenhaus Sankt Josef Braunau, Braunau am Inn
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Landeskrankenhaus Hochsteiermark, Leoben
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landeskrankenhaus Rankweil, Rankweil
  - Landeskrankenhaus Salzburg, Salzburg
  - Kardinal Schwarzenbergsches Krankenhaus, Schwarzach im Pongau
  - Landeskrankenhaus Steyr, Steyr
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Landesklinikum Waidhofen an der Ybbs, Waidhofen an der Ybbs
  - Klinikum Wels - Grieskirchen GmbH, Wels
  - Krankenhaus Wiener Neustadt, Wiener Neustadt
- Belgium (12):
  - Imelda Ziekenhuis Vzw, Bonheiden
  - Hopital Delta, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Algemeen Ziekenhuis Sint-Dimpna, Geel
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - Centres Hospitaliers Jolimont - Hopital de Jolimont, Haine Saint Paul - La Louviere
  - Jan Yperman Ziekenhuis, Ieper
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Algemeen Ziekenhuis Nikolaas Campus Sint-Niklaas, Sint-Niklaas
  - Centre Hospitalier Wallonie Picarde - site imc, Tournai
  - Centre Hospitalier Regional Verviers, Verviers
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment Alexandrovska, Sofia
  - University Multiprofile Hospital for Active Treatment Sveti Ivan Rilski EAD, Sofia
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia
  - Specialized Hospital for Active Treatment of Hematology Diseases EAD, Sofia
- Czechia (4):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Plzen, Pilsen
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (15):
  - Centre Hospitalier Rene Dubos, Amiens
  - Centre Hospitalier Henri Duffaut, Avignon
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Hopital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier Regional Universitaire de Limoges - Hopital Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Montpellier - Hopital Saint Eloi, Montpellier
  - Groupe Hospitalo Universitaire de Nimes - Hopital Caremeau, Nîmes
  - Hopital Pitie-Salpetriere, Paris
  - HÃ´pital Cochin, Paris
  - Groupe Hospitalier Necker - Enfants Malades, Paris
  - Centre Hospitalier Universitaire de Poitiers - Hopital la Miletrie, Poitiers
  - Centre Hospitalier Universitaire de Reims - Hopital Robert Debre, Reims
  - Centre Hospitalier de Saint Quentin, Saint-Quentin
  - Clinique Sainte Anne, Strasbourg
- Greece (17):
  - University General Hospital of Evros-Alexandroupolis District, Alexandroupoli
  - General Hospital Evangelismos, Athens
  - Errikos Dunant Hospital Center, Athens
  - General Hospital of Athens Georgios Gennimatas, Athens
  - General Hospital of Athens Laiko, Athens
  - Laikon University Hospital, Athens
  - University of Athens School of Medicine Alexandra Hospital, Athens
  - University General Hospital Attikon, Athens
  - Metropolitan General, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Larissa, Larissa
  - General Hospital of Patras Agios Andreas, Pátrai
  - General University Hospital of Patras Panagia i Voithia, Pátrai
  - Special Anticancer Hospital of Piraeus Metaxa, Piraeus
  - Theagenion Cancer Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki Georgios Papanikolaou, Thessaloniki
- Israel (2):
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (29):
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Unita Sanitaria Locale Toscana Centro, Bagno A Ripoli (FI)
  - Ospedale Monsignor Raffaele Dimiccoli, Barletta
  - Azienda Ospedaliera G Rummo, Benevento
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Presidio Ospedaliero Di Summa Perrino, Brindisi
  - Azienda Ospedaliera Brotzu Presidio Ospedaliero A Businco Centro di Riferimento Oncologico Regionale, Cagliari
  - Azienda Ospedaliera Santa Croce e Carle, Cuneo
  - Azienda Ospedaliera di Alessandro Manzoni Lecco, Lecco
  - Spedali Riuniti di Livorno, Livorno
  - Azienda Ospedaliera Papardo, Messina
  - IRCCS Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Presidio Ospedaliero Andrea Tortora, Pagani (SA)
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Ospedale Civile Spirito Santo, Pescara
  - Azienda Ospedaliera San Carlo, Potenza
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli, Reggio Calabria
  - Azienda Unita Sanitaria Locale Istituto di Ricovero di Reggio Emilia Arcispedale Santa Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Tor Vergata, Roma
  - Ospedale Sant Eugenio, Roma
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - Azienda Ospedaliera Sant Andrea, Roma
  - Azienda Ospedaliera Universitaria Ospedale San Giovanni di Dio e Ruggi D Aragona, Salerno
  - Presidio Ospedaliero San Giuseppe Moscati, Taranto
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino Ospedale Molinette, Torino
  - Azienda Ospedaliero Universitaria Integrata di Udine, Udine
  - Azienda Ospedaliera Universitaria Integrata di Verona Ospedale G B Rossi Borgo Roma, Verona
- Netherlands (6):
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia Ziekenhuis, locatie Langendijk, Breda
  - Sint Antonius Ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Franciscus Vlietland, Schiedam
  - HagaZiekenhuis, locatie Leyweg, The Hague
  - VieCuri Medisch Centrum, Venlo
- Oslo Universitetssykehus HF, Oslo, Norway
- Romania (12):
  - Spitalul Judetean de Urgenta Dr Constantin Opris Baia Mare, Baia Mare
  - Policlinica de Diagnostic Rapid, Brasov
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carola Davila", Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Coltea Clinical Hospital, Bucharest
  - Profesor Dr Ion Chiricuta Institut of Oncology, Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
  - Iasi Regional Oncology Institute, Iași
  - Spitalul Clinic Dr Gavril Curteanu Oradea, Oradea
  - Targu-Mures County Emergency Clinical Hospital, Târgu Mureş
  - SC Oncomed SRL, Timișoara

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Leleu X, Katodritou E, Kuehr T, Terpos E, Caers J, Zambello R, Brescianini A, Liang T, Wetten S, Badelita SN. Real-world use of carfilzomib combined with lenalidomide and dexamethasone in patients with multiple myeloma in Europe and Israel. EJHaem. 2022 Nov 6;4(1):174-183. doi: 10.1002/jha2.595. eCollection 2023 Feb. PMID 36819146
- [Background] Terpos E, Zambello R, Leleu X, Kuehr T, Badelita SN, Katodritou E, Brescianini A, Liang T, Wetten S, Caers J. Real-World Use and Effectiveness of Carfilzomib Plus Dexamethasone in Relapsed/Refractory Multiple Myeloma in Europe. Cancers (Basel). 2022 Oct 28;14(21):5311. doi: 10.3390/cancers14215311. PMID 36358731
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com